CLINICAL TRIAL: NCT02987114
Title: A Phase II, Open-label, Single-center Clinical Study to Evaluate the Safety, Tolerability and Efficacy of Oral Administration of PTL101 (Cannabidiol) as an Adjunctive Treatment for Pediatric Intractable Epilepsy
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of Oral Administration of PTL101 (Cannabidiol) as an Adjunctive Treatment for Pediatric Intractable Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoTech Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-100
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLT101 (Experimental): PTL101 capsules (50 or 100 mg CBD per capsule) up to 25 mg/kg/day or up to 450 mg/day, the lower of the two. Twice daily (morning and evening).
  Interventions: Drug: PLT101

INTERVENTIONS:
Drug: PLT101 — PTL 101 (Cannabidiol, CBD) Two piece hard capsules filled with seamless gelatin matrix green beads containing CBD (50 or 100 mg CBD per capsule) The beads should be administered following a meal, mixed with food

SUMMARY:
To evaluate the safety, tolerability and efficacy of oral administration of PTL101 (cannabidiol) for the treatment for pediatric intractable epilepsy.

Study will include a 4-week observation period ,12 weeks of treatment and 2 weeks of follow up.

DETAILED DESCRIPTION:
This is an open-label, single-center study recruiting approximately 15 male or female pediatric (ages 2-15, inclusive) patients with, intractable epilepsy, on stable doses of antiepileptic drugs (AEDs). The study comprised of the following period: 4 weeks observation period, followed by a 2-week dose titration period, 10-week maintenance treatment period, and a 2-week follow-up of which 1 week is a tapering-off period. Seizures will be recorded by the legal guardian/caregiver in seizure diaries throughout the first 16 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects with refractory epilepsy
2. 2-15 years old (inclusive), male or female
3. History of the any of the following seizure types: tonic, clonic, tonic-clonic in the form of partial seizures, partial seizures secondarily generalized or primary generalized, complex partial seizures and drop attacks (tonic/atonic).
4. At least four clinically countable seizures within 4 weeks of study entry [tonic, clonic, tonic-clonic in the form of partial seizures, partial seizures secondarily generalized or primary generalized and/or complex partial seizures and drop attacks (tonic/atonic)]
5. Subject on a stable regimen of 1-4 concomitant antiepileptic drugs (AEDs) for a minimum of 4 weeks prior to enrollment
6. History of treatment with at least four AEDs, including one trial of a combination of two concomitant drugs, without successful seizure control
7. Subjects with vagal nerve stimulation system must be on stable settings for a minimum of 6 months prior to enrollment
8. For subjects undergoing dietary treatment (e.g., ketogenic or modified Atkins diet):

   the fat to carbohydrate ratio must be stable for a minimum of eight weeks prior to enrollment
9. The subject's legal guardian voluntarily provides consent for participation in the study and signs an Informed Consent Form
10. Completed seizures diary for four weeks (±3 days) prior to initiation of the dose titration period (visit 2). Subject will be considered a screen failure if seizures diary was not appropriately completed.

Exclusion Criteria:

1. The subject is currently using or has used cannabis-based or synthetic cannabinoid within three months of study entry
2. Subject is unwilling to abstain from use of cannabis-based or synthetic cannabinoid throughout the study period
3. Neurodegenerative or deteriorated neurological disease
4. History of heart failure
5. Known family history (first-degree) of psychiatric disorders
6. Psychosis or past psychotic event and/or anxiety disorder
7. Current or history of drug abuse/addiction
8. Renal, hepatic (ALT/AST >2x upper limit of normal (ULN), bilirubin >2x ULN), pancreatic dysfunctions or laboratory test abnormalities, at the investigator's discretion
9. Clinically significant finding in baseline ECG
10. Initiation of felbamate treatment within 9 months of screening
11. Allergy to CBD or any cannabinoid and/or formulation excipients
12. Subject is pregnant, lactating, or planning a pregnancy during the course of the study or within 3 months of study completion
13. Subject and legal guardian/caregiver unable to comply with study visits/requirements
14. Subject is currently enrolled in, or has not yet completed a period of at least 60 days since ending another investigational device or drug trial(s)

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence of study treatment related adverse events (AEs) | 12 weeks of treatment + 2 weeks follow up
Percent change in mean countable monthly seizure frequency | 12 week treatment period

SECONDARY OUTCOMES:
Incidence of all adverse events (AEs) | 12 weeks of treatment + 2 weeks follow up
assessment of Caregiver Global Impression of Improvement using a 5-point rating scale | after 5 weeks of maintenance dose and at end of treatment
assessment of Caregiver Global Impression of Seizure Severity using a 5-point rating scale | after 5 weeks of maintenance dose and at end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Epilepsy department- Souraskey Medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No